CLINICAL TRIAL: NCT02347618
Title: Pilot Study of Short-Course Preoperative Stereotactic Body Radiation Therapy for Resectable Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Alan Katz, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UGIP14107
Record Dates: First submitted 2014-12-24; First posted 2015-01-27 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Pancreatic Cancer; Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative SBRT (Experimental): This will be a Phase 2, single center, prospective, single arm feasibility study of the use of stereotactic body radiotherapy (SBRT) for the preoperative treatment of surgically resectable pancreatic adenocarcinoma.
  Interventions: Radiation: Preoperative SBRT

INTERVENTIONS:
Radiation: Preoperative SBRT — This will be a Phase 2, single center, prospective, single arm feasibility study of the use of stereotactic body radiotherapy (SBRT) for the preoperative treatment of surgically resectable pancreatic adenocarcinoma.

SUMMARY:
The purpose of this study is to determine whether a short-course of stereotactic body radiotherapy (SBRT) prior to surgical resection of pancreatic adenocarcinoma is feasible and well-tolerated.

DETAILED DESCRIPTION:
This will be a Phase 2, single center, prospective, single arm feasibility study of the use of stereotactic body radiotherapy (SBRT) for the preoperative treatment of surgically resectable pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with pathologically proven diagnosis of adenocarcinoma of the head of the pancreas
2. CT w/ contrast using the pancreas protocol or MRI of the abdomen with contrast within 6 weeks prior to registration
3. CT chest or PET/CT within 6 weeks prior to registration
4. Clinically determined to be resectable based on NCCN Criteria:
5. No radiographic evidence of superior mesenteric vein or portal vein distortion
6. No evidence of distant metastasis
7. Clear fat planes around the celiac axis, hepatic artery, and superior mesenteric artery
8. No enlarged lymph nodes per CT criteria or PET avid lymph nodes
9. No lymphadenopathy outside the surgical field (i.e. celiac or para-aortic adenopathy)
10. Adequate cardiopulmonary reserves to tolerate surgery
11. Karnofsky performance status > 70
12. Age >18
13. Adequate bone marrow function defined as follows:
14. Absolute neutrophil count (ANC) > 1800 cells/mm3
15. Platelets ≥ 100,000 cells/mm3
16. Hemoglobin > 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb > 8 g/dl is acceptable.)
17. Pregnancy test must be negative for women of childbearing potential within 7 days prior to study entry
18. Patient must sign study specific informed consent prior to study entry

Exclusion Criteria:

1. Prior surgical resection of any pancreatic malignancy
2. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
3. Any prior chemotherapy or radiation for treatment of the patient's pancreatic tumor.
4. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
5. Severe, active comorbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 12 months
   2. Transmural myocardial infarction within the last 6 months
   3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration.
6. Severe, uncorrectable hepatic insufficiency and/or coagulation defects due to liver failure
7. Any evidence of distant metastases (M1)
8. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-12; Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 2 or greater toxicity | 2 years
  Number of incidence of grade 2 or greater toxicity

SECONDARY OUTCOMES:
Number of Participants with no further growth of cancer at original site (Local control) | 2 years
  Count subjects with no further growth of cancer at original site.
Count subjects with Recurrence of cancer in other body sites | 2 years
  Compare recurrence locations of treated patients relative to historical controls.
Time to Progression of pancreatic cancer | 4 years
  Duration of progression free survival of treated patients
Time to death | 4 years
  Measure duration of survival of treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Alan W Katz, MD MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT02347618/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT02347618/ICF_001.pdf